CLINICAL TRIAL: NCT02251509
Title: Rate Control in Atrial Fibrillation: A Randomized, Double-Blind, Crossover Comparison of Carvedilol and Metoprolol Tartrate
Brief Title: Rate Control in Atrial Fibrillation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 624918
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Carvedilol; Metoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol (Experimental): carvedilol BID for 2 weeks
  Interventions: Drug: Carvedilol
- Metoprolol tartrate (Experimental): Metoprolol tartrate BID for 2 weeks
  Interventions: Drug: Metoprolol tartrate

INTERVENTIONS:
Drug: Carvedilol
  Other Names: Coreg
  Arms: Carvedilol
Drug: Metoprolol tartrate
  Other Names: Lopressor
  Arms: Metoprolol tartrate

SUMMARY:
This study will evaluate the efficacy of metoprolol tartrate compared to carvedilol on heart rate control in patients with atrial fibrillation and a rapid ventricular rate.

ELIGIBILITY:
Inclusion Criteria:

* Permanent atrial fibrillation
* Baseline ventricular rate (prior to treatment) > 110 bpm

Exclusion Criteria:

* History of accessory tract re-entry tachycardia
* Ejection fraction < 35% or history of NYHA Class III/IV stage C/D heart failure
* Acute coronary syndrome, percutaneous coronary intervention, or cardiac surgery in the past 2 months
* Child-Pugh class B or C hepatic dysfunction
* Uncontrolled hypertension
* Thyroid disease
* Intolerance to beta-blockers
* History of lung disease resulting in hospitalization in the past year

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Resting heart rate | 2 weeks
  Resting heart rate less than 80 bpm

CONTACTS AND LOCATIONS:
Overall Officials: Pallavi Bellamkonda, MBBS, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States